CLINICAL TRIAL: NCT04761588
Title: An Acceptability Study to Evaluate the Adherence, Tolerance and Metabolic Control of Patients With Tyrosinaemia When Using TYR Sphere (a Food for Special Medical Purposes) as Part of Dietary Management.
Brief Title: Evaluation of TYR Sphere in France
Acronym: TYR sphere Fra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TyrSph-2020-10-16; SI 21.01.06.74121 (Other: CPP Est I); 2021-A01263-38 (Other: REC)
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Tyrosinemia; AKU
Keywords: Tyrosinemia; AKU; Alkaptonuria; Tyr Sphere; FSMP; Food for special medical purposes
MeSH Terms: conditions — Tyrosinemias; Alkaptonuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tyr sphere (Experimental): All patients to receive Tyr sphere as part of their dietary management for tyrosinaemia or alkaptonuria (AKU).
  Interventions: Dietary Supplement: Tyr sphere

INTERVENTIONS:
Dietary Supplement: Tyr sphere — Tyr sphere is a powdered, low phenylalanine and tyrosine protein substitute, containing a balanced mix of casein glycomacropeptide (cGMP) isolate, essential and non-essential amino acids, carbohydrate, fat, vitamins, minerals and the long chain polyunsaturated fatty acid (LCP) and docosahexaenoic acid (DHA). It contains sugars and sweetener.
  The product is designed to be prescribed based on its protein content, not its energy content.

SUMMARY:
10 participants aged 3 years and over with tyrosinaemia or alkaptonuria will be prescribed Tyr sphere following an assessment of their individual needs by their dietitian.

All participants will enter a 4-week evaluation period, assessing adherence and gastrointestinal tolerance. Evaluations of Tyr sphere's palatability are made at the end of the evaluation period. Dried blood spots are taken on days 1 and 28 and once per week in between.

Participants who continue to take the product at the end of their evaluation period will enter a follow-up period during which metabolic control, anthropometric and nutritional status data will be collected during the yearly standard of care routine visits.

DETAILED DESCRIPTION:
10 participants with tyrosinaemia or alkaptonuria will be invited to participate in this study. Following consent they will be assessed by their dietitian and a recommended amount of Tyr sphere will be prescribed based on their individual needs. Tyr sphere is a food for special medical purposes as defined by Regulation (EU) No 609/2013. It is designed to be prescribed based on its protein content, not its energy content.

Visit 1, baseline clinic visit activities: consent, demographics, anthropometric measurements, gastrointestinal history, dietary assessment, metabolic control assessment including collection of dried blood spots for phenylalanine and tyrosine levels, record routinely taken urine succinylacetone, serum albumin and pre-albumin levels, new dietary prescription.

Weeks 1 to 4 (patient at home): dried blood spots, adverse events reporting/assessment, daily Tyr sphere adherence diary, daily gastrointestinal symptoms diary (weeks 1 and 4 only), daily intake diary for Nitisinone which is routinely prescribed. There will be a telephone call

Visit 2, end of acceptability phase clinic visit activities: anthropometric measurements, review of diaries, review of adverse events, metabolic control assessment including collection of dried blood spots for phenylalanine and tyrosine levels, investigator's assessment of Tyr sphere for the participant and decision on continuing with the prescription.

Three-year routine follow-up: for the participants that do continue with the Tyr sphere prescription (in consultation with the investigator), they will enter a follow-up period of three years, during which only routine, standard of care visits and procedures will take place. Data will be collected on anthropometrics, phenylalanine and tyrosine levels from dried blood spots, adverse events, record routinely taken urine succinylacetone, serum albumin and pre-albumin levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with tyrosinaemia.
* Aged ≥ 3 years.
* In the opinion of the Investigator, can comply with the study protocol and take at least one sachet of the study product per day.
* Willingly given, written, informed consent from patient or parent/guardian.
* Willingly given, written assent (if appropriate).

Exclusion Criteria:

* Individuals who are allergic to milk, fish and soya (these allergens are inherent in the study product ingredients).
* Use of additional macro/micronutrient supplements during the evaluation period, unless clinically indicated and prescribed by the Investigator (must be recorded in patient case report form CRF).
* Women who are pregnant / breastfeeding at the start of the study or planning to become pregnant during the study.

N.B.: Women who become pregnant during the study will no longer be able to participate and will be withdrawn.

* Individuals who, in the opinion of the investigator, are unable to comply with the requirements of the protocol.
* Any co-morbidity, which, in the opinion of the Investigator, would preclude participation in the study.
* Patients who are currently participating in, plan to participate in, or have participated in an interventional investigational drug, food or medical device trial within 30 days prior to screening visit.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change in adherence to recommended amounts of Tyr sphere | Recorded daily on days 1-28
  Patient reported data on actual compared to prescribed intakes of Tyr sphere, assessed by HCPs periodically as per routine practice.
Change in gastrointestinal tolerance | Recorded daily on days 1-28
  Patient reported data on any gastrointestinal symptoms experienced, assessed by HCPs periodically as per routine practice.
Patient evaluation of Tyr sphere's palatability | Day 28, end of acceptability phase
  Patient-reported assessment of Tyr sphere's palatability on a Likert scale: 1 (really didn't like it) to 5 (loved it).
Change in metabolic control: tyrosine levels | Day 1, week 1, week 2, week 3, week 4, day 28
  Tyrosine levels obtained from dried blood spots
Change in metabolic control: phenylalanine levels | Day 1, week 1, week 2, week 3, week 4, day 28
  Phenylalanine levels obtained from dried blood spots

SECONDARY OUTCOMES:
Long term change in growth | 3-year follow-up period
  Recorded progress in growth from standard of care follow-up visits for three years
Long term change in urine succinylacetone level | 3-year follow-up period
  Recorded changes in urine succinylacetone levels from standard of care follow-up visits for three years
Long term change in pre-albumin level | 3-year follow-up period
  Recorded changes in pre-albumin levels from standard of care follow-up visits for three years
Long term change in serum albumin level | 3-year follow-up period
  Recorded changes in serum albumin levels from standard of care follow-up visits for three years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Arnoux, Principal Investigator — Hopital Necker-Enfants Malades
Locations (1):
- Hopital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No